CLINICAL TRIAL: NCT07282795
Title: Post-marketing Surveillance Study for the Safety of Efluelda® Pre-filled Syringe, a High-dose Trivalent Influenza Vaccine Administered to Adults 65 Years or Older in the Republic of Korea
Brief Title: Post-marketing Surveillance Study for the Safety of Efluelda® Pre-filled Syringe
Status: Not yet recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: FIM00018; U1111-1331-8205 (Registry Identifier: ICTRP)
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Influenza Immunization; Healthy Volunteers
Keywords: Flu; Efluelda®
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Efluelda® Vaccination Group: Adults aged 65 years of age or older will receive 1 dose of Efluelda® vaccination intramuscularly on Day 1
  Interventions: Biological: Efluelda® Pre-filled syringe

INTERVENTIONS:
Biological: Efluelda® Pre-filled syringe — Pharmaceutical Form:
  Suspension for injection in a pre-filled syringe Route of Administration: Intramuscular administration

SUMMARY:
To objective of this study is to investigate the incidence of adverse events (AEs) and adverse drug reactions (ADRs) occurred following administration of Efluelda® in adults aged 65 years or older under routine clinical practice, as per approved indications This is an open-label, multi-center, observational active safety surveillance study, designed to be conducted under standard healthcare setting of the Republic of Korea, in accordance with "Regulation on the Operation of Risk Management Plans".

The study duration of each participation will be approximately 28 to 35 days. In the event that Visit 2 is not made, the study duration would be extended to 36 to 42 days.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 65 years or older on the day of enrollment
* The informed consent form has been signed and dated
* Receipt of 1 dose of Efluelda® on the day of enrollment according to the approved local product label

Note: The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Exclusion Criteria:

* Previous history of enrollment in this study
* Participation at the time of study enrollment (or in the 4 weeks preceding the enrollment) or planned participation during the present study period in a clinical study investigating a vaccine, drug, medical device or medical procedure

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Investigators will recruit participants after vaccination with Efluelda® as per routine healthcare visits and according to approved local product labeling, at study centers (general hospitals or clinics located in South Korea).
  600 evaluable participants will be included and will include male and female adults aged 65 years and older.
Sampling Method: Non-Probability Sample
Enrollment: 670 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2029-02-22 (Estimated); Study Completion 2029-03-20 (Estimated)

PRIMARY OUTCOMES:
Occurrence of solicited injected site reactions. | Up to 7 days after vaccination
  Number of participants experiencing solicited injection site reactions
Occurrence of solicited systemic reactions | Up to 7 days after vaccination
  Number of participants experiencing solicited systemic reactions
Occurrence of unsolicited Adverse Events (AE) | From vaccination to Visit 2 (up to approximately 42 days)
  Number of participants experiencing AEs
Occurrence of unsolicited Adverse Drug Reactions (ADR) | From vaccination to Visit 2 (up to approximately 42 days)
  Number of participants experiencing ADRs
Occurrence of unexpected Adverse Events (AE) | From vaccination to participant's last contact (up to approximately 42 days)
  Number of participants experiencing unexpected AEs
Occurrence of unexpected Adverse Drug Reactions (ADR) | From vaccination to participant's last contact (up to approximately 42 days)
  Number of participants experiencing unexpected ADRs
Occurrence of Serious Adverse Events (SAE) | From vaccination to participant's last contact (up to approximately 42 days)
  Number of participants experiencing SAEs
Occurrence of unexpected Serious Adverse Drug Reactions (SADR) | From vaccination to participant's last contact (up to approximately 42 days)
  Number of participants experiencing unexpected SADRs
Occurrence of Adverse Event of Special Interest (AESI) | From vaccination to participant's last contact (up to approximately 42 days)
  Number of participants experiencing AESIs

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org